CLINICAL TRIAL: NCT02877862
Title: Mobile Phone Technology to Increase Genetic Counseling for Women With Ovarian Cancer and Their Families
Brief Title: Mobile Phone Technology to Increase Genetic Counseling
Acronym: mAGIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC
Record Dates: First submitted 2016-03-24; First posted 2016-08-24 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Receive 7-day mAGIC app intervention and handout
  Interventions: Behavioral: mAGIC app
- Control (No Intervention): Handout only

INTERVENTIONS:
Behavioral: mAGIC app — 7-day app to encourage uptake of genetic counseling
  Arms: Intervention

SUMMARY:
This innovative project seeks to harness mobile phone technology as a means to take preventive health care to a new level among ovarian cancer survivors. Using the Fogg Behavioral Model, developed from the concept of persuasive technology, this study proposes to develop the Mobile Application for Genetic Information on Cancer (mAGIC) intervention to motivate ovarian cancer survivors to undergo genetic counseling. The overall study objective is to develop and assess the feasibility and effectiveness of a theory-based intervention aimed to encourage ovarian cancer survivors to receive genetic counseling

DETAILED DESCRIPTION:
This project seeks to harness mobile phone technology as a means to take preventive health care to a new level among ovarian cancer survivors. Using the Fogg Behavioral Model31 (FBM), developed from the concept of persuasive technology, this study proposes to develop the Mobile Application for Genetic Information on Cancer (mAGIC) week-long intervention to motivate ovarian cancer survivors to undergo genetic counseling.

ELIGIBILITY:
Inclusion Criteria:

* Woman diagnosed with ovarian, primary peritoneal or fallopian tube cancer
* 18 years old or older
* At least a fifth grade education
* Able to read and write in English
* Voluntary written informed consent before study entry, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

• Known major psychiatric or neurological diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Uptake of cancer genetic counseling | 3 months
  Report of attendance of an appointment with genetic counselor to discuss cancer genetics related to ovarian cancer diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Geller, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vogel RI, Niendorf K, Petzel S, Lee H, Teoh D, Blaes AH, Argenta P, Rivard C, Winterhoff B, Lee HY, Geller MA. A patient-centered mobile health application to motivate use of genetic counseling among women with ovarian cancer: A pilot randomized controlled trial. Gynecol Oncol. 2019 Apr;153(1):100-107. doi: 10.1016/j.ygyno.2019.01.019. Epub 2019 Feb 1. PMID 30718125